CLINICAL TRIAL: NCT03406130
Title: Localized Piezoelectric Alveolar Decortication With Customized Orthodontic Treatment in Adults: A Randomized Controlled Trial
Brief Title: Localized Piezoelectric Alveolar Decortication With Customized Orthodontic Treatment in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: ACTEON Group (Industry)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Prof. France Lambert, University of Liege
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: P2016-1 WP1
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Tooth Overcrowding
MeSH Terms: interventions — Orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insignia orthodontic treatment (Active Comparator)
  Interventions: Procedure: Orthodontic Procedure
- Piezocision-assisted Insignia orthodontic treatment (Experimental)
  Interventions: Procedure: Orthodontic Procedure; Procedure: Piezocision surgery

INTERVENTIONS:
Procedure: Orthodontic Procedure — Damon self-ligating systems (Ormco) were used for all patients. The patients were allowed to choose between clear and metal brackets. The bonding method was standardized and applied according to the manufacturer's instructions. After bracket bonding, 0.014-in. copper nickel-titanium Damon arch forms were placed. The subjects returned every 2 wk, and the archwires were changed only when full bracket engagement were achieved. The sequence of archwires was the following: 0.018-in., 0.014 × 0.025-in., and 0.018 × 0.025-in. copper nickel-titanium archwires were used for alignment, while 0.019 × 0.025-in. stainless-steel archwires were used for fine-tuning. Following the alignment steps, impressions were taken, and a blinded senior orthodontist validated appliance removal or provided advice regarding further adjustments.
  Alginate impressions were taken after the removal of the appliances, and fixed and removable retainers were placed.
Procedure: Piezocision surgery — The piezocision surgery was performed 1 week after orthodontic appliance placement. The surgical protocol was performed as described by Dibart and al. (Dibart et al. 2009). However, to avoid bias, hard and soft tissue augmentations were not considered. The patients received local anesthesia in both arches; vertical interproximal microincisions were created below each interdental papilla. In cases of root proximity (i.e., <2 mm of interdental bone), this procedure was not performed. These incisions were kept to a minimum (varying from 5 to 8 mm). Next, with a vertical piezoelectric device, 5-mm-long and 3-mm-deep corticotomies were made, and no subsequent sutures were required. The patients were advised to take analgesics (paracetamol) only if necessary and to record their daily intake for 1 wk. Anti-inflammatories were prohibited to avoid interference with the RAP.
  Arms: Piezocision-assisted Insignia orthodontic treatment

SUMMARY:
The aim of the present randomized controlled clinical trial will compare Insignia orthodontic treatment to piezocision-assisted Insignia orthodontics in adult patients. The primary objective will be to determine the efficacy of piezocision-accelerated orthodontic treatment by measuring the treatment duration in both groups. The secondary objectives will be to compare periodontal health, alveolar crest changes, bone and gingival healing, analgesic intake and patient-centered outcomes between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring maxillary and mandible orthodontic treatment (both arches)
* Adult patients with completed growth based on the cervical vertebral maturation method as described by Baccetti et al. (Baccetti et al. 2002)
* Minimal to moderate maxillary and mandibular anterior crowding at baseline (irregularity index <6;(Little 1975));
* American Society of Anesthesiology I or II (I = nor- mal healthy patient; II = patient with mild systemic disease);
* Adequate dento-oral health (i.e., the absence of periodontal diseases, periapical infection, or untreated caries).

Exclusion Criteria:

* controlled periodontitis with a loss of alveolar support >10%
* gingival recession >2 mm
* smokers
* altered bone metabolism (e.g., due to antiresorptive drug, steroid, or immunosuppressant use)
* mental or motor disabilities; and 6) pregnancy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Overall treatment time measurement (in days) | 1 year
  The cumulative times from bracket placement to each archwire change and to orthodontic appliance removal will be recorded in days.

SECONDARY OUTCOMES:
Comparison of periodontal parameters between the test group and the control group before (at baseline) and after orthodontic treatment. | baseline, 1 year
Alveolar crest parameters measurements (CBCT in millimeters) | baseline, 1 year
  The patients will be undergone baseline and post- treatment CBCT. The thick- ness of the buccal alveolar plate and the buccolingual thickness of the alveolar crest will be measured.
Comparison of radiographic parameters between the test group and the control group before (at baseline) and after orthodontic treatment (CBCT) | baseline, 1 year
Comparison of Patient-centered outcomes (VAS questionnaire) between the test group and the control group before (at baseline) and after orthodontic treatment | baseline, 1 year

REFERENCES:
- [Derived] Charavet C, Lecloux G, Jackers N, Maes N, Lambert F. Patient-reported outcomes measures (PROMs) following a piezocision-assisted versus conventional orthodontic treatments: a randomized controlled trial in adults. Clin Oral Investig. 2019 Dec;23(12):4355-4363. doi: 10.1007/s00784-019-02887-z. Epub 2019 Apr 6. PMID 30955096
- [Derived] Charavet C, Lecloux G, Jackers N, Albert A, Lambert F. Piezocision-assisted orthodontic treatment using CAD/CAM customized orthodontic appliances: a randomized controlled trial in adults. Eur J Orthod. 2019 Sep 21;41(5):495-501. doi: 10.1093/ejo/cjy082. PMID 30649257